CLINICAL TRIAL: NCT07198425
Title: Predicting Success of Decannulation Using Wearable-derived Physiology : A Prospective Cohort Study
Brief Title: Predicting Success of Decannulation Using Wearable-derived Physiology
Status: Not yet recruiting | Type: Observational
Sponsor: Bin Zhang (Other)
Collaborators: Beijing Rehabilitation Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor-Investigator, Bin Zhang, Principal Investigator, Capital Medical University
Organization: Capital Medical University (Other)
Other Study IDs: 2025-bjkfyy-ppfs-ud
Record Dates: First submitted 2025-09-14; First posted 2025-09-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Tracheostomy Decannulation; Physiological Parameter
Keywords: speaking valve; Physiological Parameter; tracheostomy decannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Successful decannulation group — Patients who successfully completed the decannulation process and had their tubes removed, with no reinsertion of the tracheostomy tube or endotracheal intubation within 48 hours after decannulbation.
Other: Successful decannulation group — Patients who did not pass the decannulation process, and the multidisciplinary team advised against removal of the tracheostomy tube; or patients who passed the decannulation process and had the tracheostomy tube removed but required reinsertion of the tracheostomy tube or endotracheal intubation within 48 hours due to medical conditions.

SUMMARY:
The population included in this study consists of tracheostomy patients admitted to the pulmonary department of Beijing Rehabilitation Hospital, undergoing decannulation rehabilitation treatment. Once patient conditions stabilized, they were all transitioned to the decannulation process established by our department in 2018, which utilizes a speaking valve instead of capping. Physiological monitoring was performed for each enrolled patient on the day before their first use of the speaking valve, with continuous monitoring lasting 24 hours. Differences in the 24-hour physiological parameters with clinical parameters on the day before speaking valve use between the successful decannulation group and the failed decannulation group were compared.

Decannulation criteria: If the patient can tolerate wearing the speaking valve continuously for 4 hours (gradually increasing the duration: 30 minutes, 1 hour, 2 hours, 4 hours), and if PEF > 100 liters/min, planned removal of the tracheostomy tube can be considered.

Based on decannulation outcomes, patients were categorized into the successful decannulation group and the failed decannulation group.

Successful decannulation group: Patients who successfully completed the decannulation process and had their tubes removed, with no reinsertion of the tracheostomy tube or endotracheal intubation within 48 hours after decannulation.

Failed decannulation group: Patients who did not pass the decannulation process, and the multidisciplinary team advised against removal of the tracheostomy tube; or patients who passed the decannulation process and had the tracheostomy tube removed but required reinsertion of the tracheostomy tube or endotracheal intubation within 48 hours due to medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, non-mechanically ventilated patients.
* Tracheotomy completed, ≥48 hours since cannula placement (postoperative early edema has stabilized).
* Patient or legal representative has provided informed consent.
* Known contraindications for tracheotomy decannulation.

Exclusion Criteria:

* Recent (≤48 hours) major neck/upper airway surgery requiring avoidance of upper airway airflow impact.
* Severe consciousness disorder/delirium (RASS ≤ -3 or ≥ +2), extreme anxiety/inability to cooperate.
* Total laryngectomy or laryngo-tracheal separation.
* Oral endotracheal intubation.
* Age <18 years.
* Malignant tumor with an expected survival time ≤ 6 months.
* Patients or legal representatives unable to obtain informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pre-decannulation rehabilitation therapy for tracheotomy patients
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in physiological parameters between patients in the decannulation success and decannulation failure groups | During the 24 hours before wearing the speaking valve on the day of entering the decannulation process
  Primary endpoint: Whether "decannulation success" (binary: success/failure) is achieved within 48 hours after the first planned removal of the tracheostomy tube in tracheostomized patients.
  Primary Objectives: Comparing key physiological parameters between the successful and failed tracheostomy decannulation groups to identify objective indicators associated with successful decannulation.
  Secondary Objectives:
  1. Develop predictive models to assess the probability of successful decannulation prior to the procedure.
  2. Investigate the relationship between time-series features (e.g., circadian rhythms, volatility) and decannulation outcomes.
  3. Identify potentially modifiable physiological risk signals (e.g., nocturnal hypoxic burden, reduced heart rate variability).
  Wearable device data collection time: Within 24 hours after the patient enters the decannulation process and before the first use of a speaking valve.

CONTACTS AND LOCATIONS:
Overall Officials: Hongying Jiang, Study Chair — Beijing Rehabilitation Hospital of Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No